CLINICAL TRIAL: NCT04420000
Title: Effects of Mindfulness Therapy in Patients With Acromegaly and in Patients With Cushing's Syndrome
Brief Title: Effects of Mindfulness Therapy in Patients With Acromegaly and Cushing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: A.O. Ospedale Papa Giovanni XXIII (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-MIN-2020-16
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Patient Satisfaction
Keywords: Mindfulness; Acromgaly; Cushing; Quality Of Life
MeSH Terms: conditions — Patient Satisfaction | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients having a Mindfulness program
  Interventions: Behavioral: Mindfulness
- Control group (Placebo Comparator): Patients having a routinary managment
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness based programme
  Arms: Interventional group
Other: Control — Treatment as usual
  Arms: Control group

SUMMARY:
Randomized, multicenter, international clinical trial (one center in Barcelona and one center in Bergamo, Italy), with exploratory intention.

The main objective of the study will be to assess changes in quality of life, mood, chronic pain and sleep after the delivery of a Mindfulness program.

The secondary objectives will be: to evaluate if this program also affects blood pressure, if the changes are maintained six months after treatment and if it determines the decrease in health resources used.

The intervention group will do Mindfulness sessions according to an established protocol of 8 weeks, while the control group will follow the normal clinical routine. The Mindfulness protocol will be carried out in group sessions led by a therapist with experience in mindfulness and compassion, lasting 120 minutes, weekly, which will take place over 8 weeks.

Two separate studies will be done, one for patients with acromegaly which will be the first to take place and then another for patients with Cushing's syndrome.

DETAILED DESCRIPTION:
Sixty patients with acromegaly, (30 in Spain and 30 in Italy) and 60 patients with Cushing syndrome (30 in Spain and 30 in Italy), who are visited in the Endocrinology services of the Hospital de la Santa Creu i Sant Pau, Barcelona and Papa Giovanni XXIII in Bergamo will participate in the study.

In each center there will be 30 patients for each pathology (15 will participate in the Mindfulness intervention group and 15 will receive the usual treatment).

Inclusion criteria: 1) age between 18 and 70 years, 2) diagnosis of acromegaly, 3) diagnosis of Cushing's syndrome, 4) patients with controlled disease, 5) not currently participating in any other clinical study.

Exclusion criteria: 1) physical illnesses or comorbidity of serious mental illness that impede the practice of Mindfulness, 2) Patients who for cognitive, neurological or psychiatric reasons could not follow the sessions 3) Patients who do not accept signing the informed consent 4) Patients with Cushing's syndrome or active acromegaly, 5) Simultaneous participation in another clinical study.

Patients who meet the inclusion / exclusion criteria will be invited to participate in the study. The Patient Information Sheet (HIP) and Informed Consent (CI) will be provided. There will be three evaluation visits (pre and post intervention, and 6 months after the intervention) in which the participants must complete different questionnaires and scales. Participants will be invited to keep a daily practice log, and will be required to complete the assigned daily meditation practices for the 8-week program.

Demographic and clinical variables (collected from the medical history) will be included. Patients will also have their blood pressure taken before and after each session.

Questionnaires:

* Quality of Life: AcroQoL (patients with acromegaly), CushingQoL (patients with Cushing syndrome)
* Mood: Hospital Anxiety and Depression Scale (HADS)
* Sleep: Pittsburgh Sleep Quality Index
* Pain: McGill Pain Questionnaire
* Self Compassion Scale (SCS)
* Life satisfaction scale (SWLS)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of controlled acromegaly,
* Clinical diagnosis of controlled Cushing syndrome
* Must be able to perform Mindfulness

Exclusion Criteria:

* Psychiatric disorders
* Previous experience with Mindfulness
* Participation in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life in patients with acromegaly | Baseline, post-intervention (8 weeks)
  using the Acromegaly Quality of Life Questionnaire (AcroQoL)
Change in quality of life in patients with Cushing's syndrome | Baseline, post-intervention (8 weeks)
  using the Cushing's Quality-of-Life (CushingQOL) questionnaire

OTHER OUTCOMES:
Change in Pain in patients with acromegaly and Cushing's syndrome | Baseline, post-intervention (8 weeks)
  as evaluated using the McGill Pain Questionnaire
Change in Mood in patients with acromegaly and Cushing's syndrome | Baseline, post-intervention (8 weeks)
  as evaluate using Hospital Anxiety and Depression Scale (HADS)
Change in Sleep in patients with acromegaly and Cushing's syndrome | Baseline, post-intervention (8 weeks)
  as evaluate using Pittsburgh sleep scale
Self compassion in patients with acromegaly and Cushing's syndrome | Baseline, post-intervention (8 weeks)
  as evaluate using Self Compassion Scale (SCS)
Satisfation with life in patients with acromegaly and Cushing's syndrome | Baseline, post-intervention (8 weeks)
  as evaluate using SWLS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Resmini, MD, PhD, Principal Investigator — Ciberer and IIB Sant Pau
Locations (1):
- Resmini Eugenia, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
We'll publish the data after completing the study